CLINICAL TRIAL: NCT02141958
Title: An Adaptive Phase I Intra-patient Dose Escalation Study of Fenretinide in Adult Cystic Fibrosis Patients
Brief Title: Safety Study of Fenretinide in Adult Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elias Matouk (Other)
Responsible Party: Sponsor-Investigator, Elias Matouk, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MGU-4HPR-13-01
Record Dates: First submitted 2014-05-13; First posted 2014-05-20 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Fenretinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fenretinide (Experimental): Fenretinide will be administrated orally once per day for 21 consecutive days, in up to three treatment cycles of ascending doses, with a minimum of 7-day drug-free period between cycles. Twelve (12) patients will be on Fenretinide.
  Interventions: Drug: Fenretinide
- Placebo (Placebo Comparator): Four (4) patients will be on Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenretinide — Fenretinide oral capsules of 100mg, each selected dose being administered once daily for 21 days (treatment cycle). Up to three total daily dose levels will be assessed in the study, as follows: 100mg of Fenretinide (one capsule) for the first treatment cycle, 200mg of Fenretinide (two capsules) in the second treatment cycle, and 300mg or 400mg of Fenretinide (3 or 4 capsules) will be selected for the third treatment cycle, based on safety and PK data collected.
  Arms: Fenretinide
Drug: Placebo — A matching placebo will be used to keep the study double-blind.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ascending doses of a novel oral formulation of Fenretinide to adult cystic fibrosis (CF) patients, once-daily for 21 days (treatment cycle). This study will include up to three (3) dose levels with minimum 7 day breaks in between treatment cycles. For each dose level, blood samples will be collected for exploratory pharmacokinetic (PK) and pharmacodynamic (PD) evaluation.

DETAILED DESCRIPTION:
Patients with cystic fibrosis have an innate imbalance of essential fatty acids, with increased arachidonic acid (AA) levels, decreased docosahexanoic acid (DHA) levels, and elevated AA/DHA ratio. An increasing amount of evidence suggests that this lipid imbalance is a primary effect in CF, playing a major role in the infection-inflammation vicious cycle that leads to respiratory failure. Fenretinide, a derivative of vitamin A, was shown to correct the AA/DHA imbalance in lungs and blood plasma in specific animal model of CF, resulting in reduced lung inflammation and decrease in the severity of pulmonary infections with Pseudomonas aeruginosa.

This is a single center, randomized, double-blinded, placebo-controlled Phase 1 clinical study to evaluate the safety and tolerability of up to 3 increasing oral doses of Fenretinide compared to placebo, and to evaluate the pharmacokinetics of Fenretinide in adult CF patients chronically infected with Pseudomonas aeruginosa. A single cohort of 16 clinically stable adult patients will be randomized to either Fenretinide or placebo, in a 3:1 randomization scheme (12 active, 4 placebo).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Males or females
* 18 years and older
* Diagnosis: Patients must have a diagnosis of cystic fibrosis (positive sweat chloride test) or confirmation of two genetic mutations, one mutation on each of the two alleles of the Cystic fibrosis transmembrane conductance regulator (CFTR) gene causing Cystic Fibrosis
* Chronic cystic fibrosis lung disease with baseline Forced Exploratory Volume in one second equal or superior to 40% predicted value for age, gender and height
* Clinically stable patients will be enrolled in the study, i.e. stable at least one month after successful treatment of pulmonary exacerbation
* Chronic pulmonary Pseudomonas aeruginosa colonization and/or infection (sustained microbiological evidence from sputum for the past 6 months, prior to enrollment)
* Pancreatic function: Patient must take pancrelipase supplementation if diagnosed with pancreatic insufficiency as prescribed by a physician. Enzyme supplementation should not be modified during the trial
* Female patients should be on an effective contraceptive method during the study.

Exclusion Criteria:

* Pregnancy : due to the potential teratogenic effects of retinoids, pregnant women are NOT eligible
* Breastfeeding by study patient is NOT allowed
* Clinically abnormal renal function: Serum Creatinine > 132 micromoles/L
* Clinically abnormal liver function: Total bilirubin >1.5 x Upper Limit of the Normal range (ULN), Alanine Aminotransferase (ALT) and/or Aspartate AminoTransferase (AST) > 3 x ULN and Alkaline Phosphatase (ALP) > 2 x ULN
* Known history of a severe allergy or sensitivity to retinoids
* Presence of a cancerous tumor, active or in remission, treated or not
* Presence of nyctalopia or hemeralopia at enrolment, or any other serious retinal, ophthalmological condition (eg: retinitis pigmentosa, choroidoretinitis and xerophthalmia), including glaucoma
* Presence of serious dermatological conditions at entry, including inflammatory or xerotic pathologies such as psoriasis or ichthyosis
* Prior therapy with Fenretinide. Other retinoids (eg: vitamin A supplements) are allowed, but their dosing regimen should remain constant throughout the study
* Participation in another drug clinical trial within 30 days prior to the enrollment
* Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study
* Patients unable to comply with the study protocol and follow-up schedule for any psychological, familial, sociological or geographical reason.
* Patients with known allergies to excipients in the oral capsule formulation proposed to be used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of ascending doses of oral Fenretinide, each dose to be administered to adult cystic fibrosis (CF) patients once-daily (QD) during a 21 days treatment cycle. | During a 21 days treatment cycle, from time taking first dose (Day 1) through last day of each treatment cycle (Day 21)
  Changes in clinical signs and symptoms of safety data during a 21 days treatment cycle, such safety data assessment including physical examinations, ECGs, vital signs, pulmonary function (spirometry), clinical laboratory results, assessment of ophthalmological condition, and adverse events reported. The safety data will be used to authorize dose escalations. Up to three (3) doses of Fenretinide will be assessed in up to three (3) treatment cycles of 21 days.

SECONDARY OUTCOMES:
Pharmacokinetic profile of the drug, measuring Cmax, Tmax, T1/2, AUC (area under the curve) and Css (steady state concentration), for each dose level | Day 1 and 21 of each treatment cycle
  Cmax, Tmax, T 1/2, and Css (steady state concentration) with target plasma levels of Fenretinide 1-2 µM as a pharmacokinetic / pharmacodynamic biological activity
Pharmacodynamic lipid markers: plasma Arachidonic Acid (AA) and Docosahexaenoic Acid (DHA) | At baseline and Day 21 of each treatment cycle
  Arachidonic Acid as omega-6 proinflammatory fatty acid and Docosahexaenoic Acid (DHA) as an omega-3 anti-inflammatory fatty acid.
Pharmacodynamic inflammatory markers: Immunoglobulin G, Interleukin 1β, Interleukin 6, Interleukin 8, Interleukin 10, Macrophage inflammatory protein-1β, Tumor necrosis factors and Vascular endothelial growth factor | At baseline and Day 21 of each treatment t cycle

OTHER OUTCOMES:
Pre-specified exploratory parameter: pulmonary function using the Forced Expiratory Volume in 1 second test | At baseline and Day 21 of each treatment cycle
  Forced expired volume in 1 second as percent predicted according to age, gender and height
Pre-specified exploratory parameter: quality of life using the Cystic Fibrosis Quality of life Questionnaire Revised (CFQ-R) | At baseline and Day 21 of each treatment cycle
  respiratory symptom score, physical domain and health perception domain

CONTACTS AND LOCATIONS:
Overall Officials: Elias Matouk, MD, Principal Investigator — Montreal Chest Institute
Locations (1):
- Montreal Chest Institute, Montreal, Quebec, Canada